CLINICAL TRIAL: NCT00642278
Title: A Randomized, Double-Blind, Placebo-Controlled, Double-Dummy, Parallel Group, Multicenter, Dose-Ranging Study in Subjects With Type 2 Diabetes Mellitus to Evaluate the Efficacy, Safety, and Tolerability of Orally Administered SGLT2 Inhibitor JNJ-28431754 With Sitagliptin as a Reference Arm
Brief Title: An Efficacy, Safety, and Tolerability Study of Canagliflozin (JNJ-28431754) in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014587; 28431754DIA2001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type II; Diabetes Mellitus, Non Insulin Dependent
Keywords: Type 2 diabetes mellitus; Metformin; Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Canagliflozin 50 mg daily (Experimental): Each patient will receive 50 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Canagliflozin 100 mg daily (Experimental): Each patient will receive 100 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Canagliflozin 200 mg daily (Experimental): Each patient will receive 200 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Canagliflozin 300 mg daily (Experimental): Each patient will receive 300 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo capsule once daily (in the evening).
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo
- Canagliflozin 300 mg twice daily (Experimental): Each patient will receive 300 mg of canagliflozin (JNJ-28431754) twice daily for 12 weeks.
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Sitagliptin 100 mg daily (Active Comparator): Each patient will receive 100 mg of sitagliptin once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
  Interventions: Drug: Sitagliptin; Drug: Placebo
- Placebo (Placebo Comparator): Each patient will receive matching placebo twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin (JNJ-28431754) — One 50 mg, 100 mg, 200 mg, or 300 mg over-encapsulated tablet orally (by mouth) once daily for 12 weeks or one 300 mg over-encapsulated tablet orally twice daily for 12 weeks.
  Other Names: JNJ-28431754
  Arms: Canagliflozin 100 mg daily; Canagliflozin 200 mg daily; Canagliflozin 300 mg daily; Canagliflozin 300 mg twice daily; Canagliflozin 50 mg daily
Drug: Sitagliptin — One 100 mg over-encapsulated tablet orally (by mouth) once daily for 12 weeks.
  Arms: Sitagliptin 100 mg daily
Drug: Placebo — One matching placebo capsule orally (by mouth) once or twice daily for 12 weeks.
  Arms: Canagliflozin 100 mg daily; Canagliflozin 200 mg daily; Canagliflozin 300 mg daily; Canagliflozin 50 mg daily; Placebo; Sitagliptin 100 mg daily

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety, and tolerability of JNJ-28431754 compared with placebo in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a metabolic disorder that is characterized by decreased secretion of insulin by the pancreas and resistance to the action of insulin in various tissues (muscle, liver, and adipose), which results in impaired glucose uptake. Chronic hyperglycemia leads to progressive impairment of insulin secretion and to insulin resistance of peripheral tissues in diabetes (so-called glucose toxicity), which further worsens control of blood glucose. In addition, chronic hyperglycemia is a major risk factor for complications, including heart disease, retinopathy, nephropathy, and neuropathy. Although numerous treatments have been developed for the treatment of diabetes and individual agents may be highly effective for some patients, it is still difficult to maintain optimal glycemic control in most patients with diabetes. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter, dose-ranging study to determine the efficacy, safety and tolerability of JNJ-28431754 taken orally over 12 weeks, compared with placebo, in the treatment of Type 2 diabetes mellitus. The primary clinical hypothesis is that JNJ-28431754 is superior to placebo as measured by the change in hemoglobin A1c from baseline through Week 12 in the treatment of type 2 diabetes mellitus. Subject safety will be monitored throughout the study using spontaneous adverse event reporting, clinical laboratory tests (hematology, serum chemistry, urinalysis); severe and serious hypoglycemic episodes, assessment of urinary albumin excretion and markers of proximal renal tubular function; pregnancy tests; electrocardiograms (ECGs); vital sign measurements; physical examinations, assessment of calcium and phosphate homeostasis, bone formation and resorption markers, and hormones regulating calcium and phosphorus homeostasis; and vaginal and urine sample collection for fungal and bacterial culture in subjects with symptoms consistent with vulvovaginal candidiasis (VVC) or urinary tract infection (UTI).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of type 2 diabetes mellitus
* Hemoglobin A1c levels >=7% and <=10.5%
* taking a stable daily dose of metformin
* Body mass index (BMI) 25 to 45 kg/m2 except those of Asian descent who must have a BMI of 24 to 45 kg/m2
* Stable body weight
* Serum creatinine <=1.5 mg/dL (132.6 umol/L) for men and <=1.4 mg/dL (123.76 umol/L) for women

Exclusion Criteria:

* Patients must not have prior exposure or known contraindication or suspected hypersensitivity to canagliflozin (JNJ-28431754)
* Known contraindication or suspected hypersensitivity to sitagliptin or metformin
* A history of diabetic ketoacidosis or type 1 diabetes mellitus
* History of pancreas or beta-cell transplantation
* History of active proliferative diabetic retinopathy
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (78):
- United States (30):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Tucson, Arizona
  - Encinitas, California
  - Lincoln, California
  - Los Angeles, California
  - Merced, California
  - Roseville, California
  - Denver, Colorado
  - Golden, Colorado
  - Hollywood, Florida
  - Jacksonville, Florida
  - Boise, Idaho
  - Nampa, Idaho
  - Topeka, Kansas
  - Haverhill, Massachusetts
  - Cherry Hill, New Jersey
  - Albuquerque, New Mexico
  - New Hyde Park, New York
  - Salisbury, North Carolina
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Greer, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - New Braunfels, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Milwaukee, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Bueos Aires
- Bulgaria (2):
  - Pleven
  - Sofia
- Canada (8):
  - Chilliwack, British Columbia
  - Coquitlam, British Columbia
  - Brampton, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Pointe-Claire, Quebec
  - Saint Romuald, Quebec
  - Saskatoon, Saskatchewan
- Czechia (3):
  - Olomouc
  - Písek
  - Prague
- India (4):
  - Bangalore
  - Hyderabad
  - Nagpur
  - Pune
- Malaysia (2):
  - Kota Bharu
  - Kuala Lumpur
- Mexico (4):
  - Mexico City
  - México
  - Monterrey
  - Zapopan
- Poland (8):
  - Bydgoszcz
  - Gdansk
  - Kutno
  - Lodz
  - Lublin
  - Torun
  - Warsaw
  - Wroclaw
- Puerto Rico (2):
  - Ponce Pr
  - San Juan
- Romania (6):
  - Baia Mare
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Galati
  - Ploieşti
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Samara
- United Kingdom (4):
  - Belfast
  - Bolton
  - Exeter
  - Lincoln

REFERENCES:
- [Derived] Nyirjesy P, Zhao Y, Ways K, Usiskin K. Evaluation of vulvovaginal symptoms and Candida colonization in women with type 2 diabetes mellitus treated with canagliflozin, a sodium glucose co-transporter 2 inhibitor. Curr Med Res Opin. 2012 Jul;28(7):1173-8. doi: 10.1185/03007995.2012.697053. Epub 2012 Jun 14. PMID 22632452
- [Derived] Nicolle LE, Capuano G, Ways K, Usiskin K. Effect of canagliflozin, a sodium glucose co-transporter 2 (SGLT2) inhibitor, on bacteriuria and urinary tract infection in subjects with type 2 diabetes enrolled in a 12-week, phase 2 study. Curr Med Res Opin. 2012 Jul;28(7):1167-71. doi: 10.1185/03007995.2012.689956. Epub 2012 May 15. PMID 22548646
- [Derived] Rosenstock J, Aggarwal N, Polidori D, Zhao Y, Arbit D, Usiskin K, Capuano G, Canovatchel W; Canagliflozin DIA 2001 Study Group. Dose-ranging effects of canagliflozin, a sodium-glucose cotransporter 2 inhibitor, as add-on to metformin in subjects with type 2 diabetes. Diabetes Care. 2012 Jun;35(6):1232-8. doi: 10.2337/dc11-1926. Epub 2012 Apr 9. PMID 22492586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of canagliflozin (JNJ-28431754) in patients with type 2 diabetes mellitus with sitagliptin as a reference arm. The study was conducted between 27 March 2008 and 28 January 2009 and recruited patients from 85 study centers located in 13 countries worldwide.
Pre-assignment Details: A total of 451 patients were randomly allocated to the 7 treatment arms in the study and comprised the intent-to-treat analysis set which was used for the efficacy analyses. All 451 patients received at least 1 dose of study drug and were included in the safety analysis set.
Groups:
- Placebo: Each patient received matching placebo twice daily for 12 weeks.
- Canagliflozin 50 mg Daily: Each patient received 50 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
- Canagliflozin 100 mg Daily: Each patient received 100 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
- Canagliflozin 200 mg Daily: Each patient received 200 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
- Canagliflozin 300 mg Daily: Each patient received 300 mg of canagliflozin (JNJ-28431754) once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
- Canagliflozin 300 mg Twice Daily: Each patient received 300 mg of canagliflozin (JNJ-28431754) twice daily for 12 weeks.
- Sitagliptin 100 mg Daily: Each patient received 100 mg of sitagliptin once daily (in the morning) for 12 weeks with matching placebo once daily (in the evening).
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Started | 65 | 64 | 64 | 65 | 64 | 64 | 65
Completed | 55 | 59 | 59 | 56 | 56 | 57 | 60
Not Completed | 10 | 5 | 5 | 9 | 8 | 7 | 5
Not completed — Adverse Event | 2 | 1 | 3 | 1 | 2 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 1 | 0 | 1 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 3 | 6 | 2 | 2
Not completed — Noncompliance with study drug regimen | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily | Total
Number analyzed (Participants) | 65 | 64 | 64 | 65 | 64 | 64 | 65 | 451
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 63 | 61 | 63 | 61 | 63 | 62 | 65 | 438
  >=65 years | 2 | 3 | 1 | 4 | 1 | 2 | 0 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 53.3 (7.82) | 53.3 (8.48) | 51.7 (7.95) | 52.9 (9.56) | 52.3 (6.88) | 55.2 (7.14) | 51.7 (8.09) | 52.9 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 28 | 32 | 28 | 36 | 27 | 215
  Male | 31 | 34 | 36 | 33 | 36 | 28 | 38 | 236
Region Enroll [Number; unit: participants]
  ARGENTINA | 1 | 1 | 3 | 1 | 2 | 0 | 2 | 10
  BULGARIA | 1 | 1 | 1 | 0 | 3 | 3 | 1 | 10
  CANADA | 11 | 6 | 9 | 8 | 8 | 4 | 7 | 53
  CZECH REPUBLIC | 2 | 3 | 2 | 6 | 0 | 2 | 2 | 17
  INDIA | 4 | 6 | 3 | 5 | 2 | 6 | 4 | 30
  MALAYSIA | 3 | 0 | 6 | 2 | 4 | 1 | 3 | 19
  MEXICO | 4 | 6 | 9 | 9 | 6 | 14 | 2 | 50
  POLAND | 3 | 5 | 4 | 7 | 6 | 5 | 9 | 39
  ROMANIA | 9 | 8 | 4 | 6 | 6 | 5 | 8 | 46
  RUSSIAN FEDERATION | 5 | 7 | 5 | 2 | 6 | 3 | 4 | 32
  UNITED KINGDOM | 1 | 0 | 2 | 1 | 3 | 1 | 2 | 10
  UNITED STATES | 21 | 21 | 16 | 18 | 18 | 20 | 21 | 135

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 12
Description: The table below shows the mean change in HbA1c from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: This analysis was conducted using the intent-to-treat analysis set, which included all patients who were randomly assigned to a treatment group. The last-observation-carried-forward method was applied when Week 12 values were missing. The table includes only patients with both baseline and post baseline values.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Number analyzed (Participants) | 61 | 62 | 62 | 62 | 60 | 62 | 62
Percent | -0.22 (0.702) | -0.79 (0.749) | -0.76 (0.992) | -0.70 (0.720) | -0.92 (0.695) | -0.95 (0.704) | -0.74 (0.615)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's procedure; ANCOVA model included terms for treatment, baseline value, and stratification factor (participation in mixed meal tolerance test); Least-Squares Mean Difference = -0.45, 95% CI 2-sided [-0.747 to -0.148], Standard Error of Mean 0.116
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's procedure; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -0.51, 95% CI 2-sided [-0.804 to -0.207], Standard Error of Mean 0.116
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 200 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's procedure; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -0.54, 95% CI 2-sided [-0.841 to -0.244], Standard Error of Mean 0.116
Statistical Analysis 4: Comparison: Placebo vs Canagliflozin 300 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's procedure; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -0.71, 95% CI 2-sided [-1.006 to -0.405], Standard Error of Mean 0.117
Statistical Analysis 5: Comparison: Placebo vs Canagliflozin 300 mg Twice Daily; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's procedure; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -0.73, 95% CI 2-sided [-1.029 to -0.432], Standard Error of Mean 0.116
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 100 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's procedure; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -0.56, 95% CI 2-sided [-0.862 to -0.265], Standard Error of Mean 0.116

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 12
Description: The table below shows the mean change in FPG from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Number analyzed (Participants) | 62 | 63 | 63 | 62 | 61 | 62 | 64
mmol/L | 0.2 (1.58) | -0.9 (2.26) | -1.4 (1.70) | -1.5 (2.23) | -1.4 (1.87) | -1.3 (1.54) | -0.7 (1.77)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Daily; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -0.9, 95% CI 2-sided [-1.39 to -0.34], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -1.4, 95% CI 2-sided [-1.98 to -0.92], Standard Error of Mean 0.27
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 200 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -1.8, 95% CI 2-sided [-2.33 to -1.27], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs Canagliflozin 300 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -1.8, 95% CI 2-sided [-2.32 to -1.26], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Placebo vs Canagliflozin 300 mg Twice Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -1.7, 95% CI 2-sided [-2.25 to -1.19], Standard Error of Mean 0.27
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 100 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -1.0, 95% CI 2-sided [-1.51 to -0.46], Standard Error of Mean 0.27

3. Secondary Outcome: Percentage of Patients With Symptoms of Hypoglycemia
Description: The table below shows the percentage of patients who experienced symptomatic hypoglycemic events between Baseline and Week 12.
Time Frame: Up to Week 12
Population: This analysis was conducted using the intent-to-treat analysis set, which included all patients who were randomiy assigned to a treatment group.
Measure: Number; unit: Percentage of patients
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Number analyzed (Participants) | 65 | 64 | 64 | 65 | 64 | 64 | 65
Percentage of patients | 2 | 0 | 2 | 6 | 0 | 3 | 5

4. Secondary Outcome: Change in Overnight Urine Glucose/Creatinine Ratio From Baseline to Week 12
Description: The table below shows the mean change in overnight urine glucose/creatinine ratio from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Number analyzed (Participants) | 54 | 58 | 56 | 53 | 57 | 56 | 58
mg/mg | 1.9 (12.34) | 35.4 (28.98) | 51.5 (28.83) | 50.5 (24.38) | 49.4 (38.41) | 61.6 (37.85) | -1.9 (14.78)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = 36.1, 95% CI 2-sided [26.07 to 46.13], Standard Error of Mean 5.10
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = 49.3, 95% CI 2-sided [39.17 to 59.34], Standard Error of Mean 5.13
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 200 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = 48.2, 95% CI 2-sided [37.98 to 58.42], Standard Error of Mean 5.2
Statistical Analysis 4: Comparison: Placebo vs Canagliflozin 300 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = 49.0, 95% CI 2-sided [38.91 to 59.01], Standard Error of Mean 5.11
Statistical Analysis 5: Comparison: Placebo vs Canagliflozin 300 mg Twice Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = 60.3, 95% CI 2-sided [50.17 to 70.35], Standard Error of Mean 5.13
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 100 mg Daily; Test type: Superiority or Other; p = 0.513, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Squares Mean Difference = -3.3, 95% CI 2-sided [-13.33 to 6.67], Standard Error of Mean 5.09

5. Secondary Outcome: Absolute Change in Body Weight From Baseline to Week 12
Description: The table below shows the mean absolute change in body weight from Baseline to Week 12 for each treatment group.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Number analyzed (Participants) | 62 | 63 | 64 | 63 | 62 | 62 | 64
kg | -0.78 (2.099) | -1.96 (2.334) | -2.25 (2.145) | -2.32 (2.842) | -2.88 (2.391) | -2.87 (2.344) | -0.43 (2.693)

6. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 12
Description: The table below shows the mean percent change in body weight from Baseline to Week 12 for each treatment group. The statistical analyses show the treatment differences (ie, each canagliflozin or sitagliptin group minus placebo) in the least-squares mean change.
Time Frame: Day 1 (Baseline) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Number analyzed (Participants) | 62 | 63 | 64 | 63 | 62 | 62 | 64
Percent change | -1.1 (2.4) | -2.3 (2.8) | -2.6 (2.3) | -2.7 (3.0) | -3.4 (2.8) | -3.4 (2.6) | -0.6 (3.0)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 50 mg Daily; Test type: Superiority or Other; p = 0.009, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = -1.3, 95% CI 2-sided [-2.2 to -0.3], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Placebo vs Canagliflozin 100 mg Daily; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = -1.5, 95% CI 2-sided [-2.5 to -0.6], Standard Error of Mean 0.5
Statistical Analysis 3: Comparison: Placebo vs Canagliflozin 200 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included terms for treatment, baseline value, and mixed meal tolerance test; Least-Sqaures Mean Difference = -1.6, 95% CI 2-sided [-2.6 to -0.7], Standard Error of Mean 0.5
Statistical Analysis 4: Comparison: Placebo vs Canagliflozin 300 mg Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = -2.3, 95% CI 2-sided [-3.3 to -1.4], Standard Error of Mean 0.5
Statistical Analysis 5: Comparison: Placebo vs Canagliflozin 300 mg Twice Daily; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = -2.3, 95% CI 2-sided [-3.3 to -1.4], Standard Error of Mean 0.5
Statistical Analysis 6: Comparison: Placebo vs Sitagliptin 100 mg Daily; Test type: Superiority or Other; p = 0.371, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least-Sqaures Mean Difference = 0.4, 95% CI 2-sided [-0.5 to 1.4], Standard Error of Mean 0.5

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study; each patient participated in the study for approximately 12 weeks.
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Event" table are based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Arm/Group | Placebo | Canagliflozin 50 mg Daily | Canagliflozin 100 mg Daily | Canagliflozin 200 mg Daily | Canagliflozin 300 mg Daily | Canagliflozin 300 mg Twice Daily | Sitagliptin 100 mg Daily
Serious Adverse Events (participants affected / at risk) | 1/65 | 1/64 | 1/64 | 1/65 | 1/64 | 1/64 | 0/65
Other Adverse Events (participants affected / at risk) | 9/65 | 13/64 | 10/64 | 10/65 | 10/64 | 12/64 | 7/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Canagliflozin 50 mg Daily (N=64) | Canagliflozin 100 mg Daily (N=64) | Canagliflozin 200 mg Daily (N=65) | Canagliflozin 300 mg Daily (N=64) | Canagliflozin 300 mg Twice Daily (N=64) | Sitagliptin 100 mg Daily (N=65)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gestational diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Canagliflozin 50 mg Daily (N=64) | Canagliflozin 100 mg Daily (N=64) | Canagliflozin 200 mg Daily (N=65) | Canagliflozin 300 mg Daily (N=64) | Canagliflozin 300 mg Twice Daily (N=64) | Sitagliptin 100 mg Daily (N=65)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 3 | 5 | 1
Nasopharyngitis (Infections and infestations) | 2 | 5 | 0 | 0 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 4 | 3 | 2 | 6 | 2 | 3 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 4 | 2 | 4 | 1 | 3 | 1
Headache (Nervous system disorders) | 2 | 1 | 5 | 2 | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.